CLINICAL TRIAL: NCT05920369
Title: The Combined Effect of Extracorporeal Shock Wave and a Tailored Exercise Program on Axillary Web Syndrome After Breast Cancer Surgery With Axillary Dissection: A Comparative, Controlled Clinical Trial.
Brief Title: Extracorporeal Shock Wave and a Tailored Exercise Program on Axillary Web Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany Mohamed Ibrahim Elgohary, associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F.P.T2207006
Record Dates: First submitted 2023-06-08; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Axillary Web Syndrome
Keywords: axillary web syndrome; shock wave; exercises; breast cancer surgery
MeSH Terms: conditions — Motor Activity | interventions — tetraethylpyrazine

STUDY DESIGN:
Intervention Model Description: controlled, double-blinded, randomized clinical trial, three arms
Who Masked: Participant, Outcomes Assessor
Masking Description: a well-experienced outcome assessor and participants are blind to the assignment of groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low-energy extracorporeal shockwave and a tailored exercise program (Experimental): the patient will be positioned lying supine with the affected shoulder in an abducted position to expose the axillary cords. Each patient received a total of 3000 shocks, which were delivered to different areas, including 1000 shocks to the axillary area, 500 shocks to the upper arm, 1000 shocks along the course of the cords, and 500 shocks to the antecubital space. Extracorporeal shock wave therapy (ESWT) was administered in two sessions during the first two weeks of the intervention, and one session each in the 3rd and 4th weeks. The energy flux density was 4 Hz with a 0.056-0.068 mJ/mm range.
  in addition to the following types of exercises: Snow Angel, Butterfly Wings, Forward Pinky Slide, Corner Stretch, Chest Stretch, Self-tissue Stretching, Overhead Moose Stretch, and Crescent Side Bend exercises
  Interventions: Other: low-energy extracorporeal shockwave and a tailored exercise program; Other: low-energy extracorporeal shockwave; Other: tailored exercise program
- low-energy extracorporeal shockwave (Active Comparator): the patient will be positioned lying supine with the affected shoulder in an abducted position to expose the axillary cords. Each patient received a total of 3000 shocks, which were delivered to different areas, including 1000 shocks to the axillary area, 500 shocks to the upper arm, 1000 shocks along the course of the cords, and 500 shocks to the antecubital space. Extracorporeal shock wave therapy (ESWT) was administered in two sessions during the first two weeks of the intervention, and one session each in the 3rd and 4th weeks. The energy flux density was 4 Hz with a 0.056-0.068 mJ/mm range.
  Interventions: Other: low-energy extracorporeal shockwave
- tailored exercise program (Active Comparator): Snow Angel, Butterfly Wings, Forward Pinky Slide, Corner Stretch, Chest Stretch, Self-tissue Stretching, Overhead Moose Stretch, and Crescent Side Bend exercises. a combination of all these types of exercises will be used. Repeat these exercises 5 times, with 3 repetitions done each day for four consecutive weeks.
  Interventions: Other: tailored exercise program

INTERVENTIONS:
Other: low-energy extracorporeal shockwave and a tailored exercise program — the patient will be positioned lying supine with the affected shoulder in an abducted position to expose the axillary cords. Each patient received a total of 3000 shocks, which were delivered to different areas, including 1000 shocks to the axillary area, 500 shocks to the upper arm, 1000 shocks along the course of the cords, and 500 shocks to the antecubital space. Extracorporeal shock wave therapy (ESWT) was administered in two sessions during the first two weeks of the intervention, and one session each in the 3rd and 4th weeks. The energy flux density was 4 Hz with a range of 0.056-0.068 mJ/mm.
  Snow Angel, Butterfly Wings, Forward Pinky Slide, Corner Stretch, Chest Stretch, Self-tissue Stretching, Overhead Moose Stretch, and Crescent Side Bend exercises
  Other Names: ESWTTEP
  Arms: low-energy extracorporeal shockwave and a tailored exercise program
Other: low-energy extracorporeal shockwave — the patient will be positioned lying supine with the affected shoulder in an abducted position to expose the axillary cords. Each patient received a total of 3000 shocks, which were delivered to different areas, including 1000 shocks to the axillary area, 500 shocks to the upper arm, 1000 shocks along the course of the cords, and 500 shocks to the antecubital space. Extracorporeal shock wave therapy (ESWT) was administered in two sessions during the first two weeks of the intervention, and one session each in the 3rd and 4th weeks. The energy flux density was 4 Hz with a range of 0.056-0.068 mJ/mm.
  Other Names: ESWT
  Arms: low-energy extracorporeal shockwave; low-energy extracorporeal shockwave and a tailored exercise program
Other: tailored exercise program — Snow Angel, Butterfly Wings, Forward Pinky Slide, Corner Stretch, Chest Stretch, Self-tissue Stretching, Overhead Moose Stretch, and Crescent Side Bend exercises
  Other Names: TEP
  Arms: low-energy extracorporeal shockwave and a tailored exercise program; tailored exercise program

SUMMARY:
A total of 93 suitable patients will be randomly allocated into three groups: Group A will receive both low-energy extracorporeal shock wave therapy and a tailored exercise program, Group B will receive only low-energy extracorporeal shock wave therapy, and Group C will receive only the tailored exercise program.

DETAILED DESCRIPTION:
Patients were randomly assigned to one of three groups: Group A, which received a low-energy extracorporeal shockwave treatment and a tailored exercise program; Group B, which received only a low-energy extracorporeal shockwave treatment; and Group C, which received only the tailored exercise program. The randomization process was done using a computer-generated table of random numbers concealed by sealed opaque envelopes. The patients' shoulder range of motion, pain intensity, upper extremity activities, and echogenicity, thickness, and disorganization were assessed using a digital inclinometer, visual analogue scale, quick DASH scale, and diagnostic ultrasound, respectively. The randomization process was overseen by a professional physical therapist who was not involved in the study procedures.

All outcomes were measured at the baseline and four weeks post-intervention. The outcomes were collected by a well-experienced investigator who was blind to the group assignments and considered as part of the research team.

ELIGIBILITY:
Inclusion Criteria:

* female
* between the ages of 40 and 65 years

Exclusion Criteria:

* metastases of any kind
* lymphedema,
* a traumatic injury to the targeted upper extremity
* a musculoskeletal disorder
* taking any anticoagulants
* had undergone bilateral breast cancer surgery
* experienced locoregional recurrence
* had vascular problems in the affected upper extremity

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
digital inclinometer | 4 weeks
  digital inclinometer will be used for the assessment of the shoulder range of motion. The inclinometer is placed near the shoulder at the proximal area with the patient's feet fixed, and the patients then moves their shoulder in different directions (flexion and abduction). The examiner repeats the measurements three times and takes the mean value as the proven measurement.

SECONDARY OUTCOMES:
visual analogue scale | 4 weeks
  the visual analog scale will be used for the assessment of pain intensity. It is a 100mm horizontal continuous line that begins on the left side with no pain and ends on the right side with more pain. The visual analogue point that corresponds to the patient's level of pain was asked to be marked by the patients. The researcher determines a score between 0 and 100 mm by measuring the distance (mm) on the 10 cm line between the patient's mark and the "no pain" sign at the left side end
Quick DASH score | 4 weeks
  the Quick DASH will be used for the assessment of upper limb disability by using shoulder and hand functions. the Arabic version of the Shortened Disabilities of the Arm, Shoulder, and Hand questionnaire (Quick DASH) is a reliable and valid measure for assessing disabilities in the upper extremities of Arabic-speaking populations. Its Cronbach's alpha of 0.89 indicates good internal consistency, while its ICC of 0.94 suggests that it has good test-retest reliability
Ultrasonography | 4 weeks
  this device will be used for the assessment of axillary cord thickness, echogenecity and disorganization. One technique used in ultrasonography is utilizing a high-resolution ultrasound system with 18 MHz frequency, which provides high-definition superficial imaging. A gel technique is also used to reduce artifacts caused by tissue compression. This technique can be used to measure cord thickness, echogenicity, and disorganization

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Hany Mohamed Elgohary, Cairo
  - Mohamed, Cairo

IPD SHARING:
Plan to Share IPD: No
results

REFERENCES:
- [Background] Elgohary HM, Al Jaouni SK, Selim SA. Effect of ultrasound-enhanced Nigella sativa seeds oil on wound healing: An animal model. J Taibah Univ Med Sci. 2018 Jun 27;13(5):438-443. doi: 10.1016/j.jtumed.2018.02.008. eCollection 2018 Oct. PMID 31435359